CLINICAL TRIAL: NCT01636089
Title: Bicarbonates Versus Saline for Contrast Induced Acute Kidney Injury Prevention in Intensive Care Unit
Acronym: HYDRAREA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: 2011-A00227-34
Record Dates: First submitted 2012-02-15; First posted 2012-07-10 (Estimated); Last update posted 2015-02-03 (Estimated); Status verified 2015-02

CONDITIONS: Contrast Induced Acute Kidney Injury
Keywords: intensive care unit
MeSH Terms: interventions — Bicarbonates; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- bicarbonates (Experimental): sodium bicarbonates 1,4%
  Interventions: Drug: bicarbonates
- saline (Active Comparator): sodium chloride 0,9%
  Interventions: Drug: saline

INTERVENTIONS:
Drug: bicarbonates — sodium bicarbonates 1,4%
  Arms: bicarbonates
Drug: saline — sodium chloride 0,9%
  Arms: saline

SUMMARY:
The aim of this study is to compare bicarbonates versus saline for prevention of contrast induced acute kidney injury in critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* patient > 18 years old
* in intensive care unit since 24h and for up to 48 hours
* with contrast medium injection

Exclusion Criteria:

* patient under renal replacement therapy
* rise in creatinine > 26µmol/L within 48hours
* anuria within 12 hours
* cardiogenic pulmonary oedema
* pH > 7.50 or kaliemia < 3mmol/L
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2012-02; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
contrast induced acute kidney injury | 72 hours

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Medical Intensive Care Unit, Caen
  - Surgical Intensive Care Unit, Caen
  - Intensive care unit, Saint-Lô